CLINICAL TRIAL: NCT04673591
Title: Effects of Tregalizumab on Allergen-induced Airway Responses and Airway Inflammation in Asthmatic Patients
Acronym: Tregulaire
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: T-Balance Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OG-061-01
Record Dates: First submitted 2020-11-26; First posted 2020-12-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Allergy to House Dust Mite; Allergic Asthma
Keywords: Mild asthma; House Dust Mite; Allergy
MeSH Terms: conditions — Dust Mite Allergy; Hypersensitivity | interventions — tregalizumab

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tregalizumab (Experimental)
  Interventions: Drug: Tregalizumab
- Matched placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tregalizumab — a monoclonal antibody designed for the treatment of allergic asthma indication
  Arms: Tregalizumab
Other: Placebo — Matched Placebo
  Arms: Matched placebo

SUMMARY:
The study will be conducted as a randomized, double-blind, placebo-controlled, single-center study in adult patients with mild controlled allergic asthma and house dust mite allergy.

DETAILED DESCRIPTION:
This study will consist of a screening phase, a treatment phase and a follow-up phase.

Eligible subjects will undergo a bronchial allergen provocation (BAP) with mite allergen to assess the asthmatic response before and after treatment. Subjects will be randomized to two parallel treatment groups. Each subject will be treated weekly over 12 weeks either with test product or with the reference product (placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent.
2. Male or female subject aged 18 to 65 years (both inclusive).
3. Established diagnosis of mild controlled allergic asthma (GINA 2019) and history of allergic bronchial asthma for at least 1 year.
4. BMI of 18.0 to 30.0 (both inclusive).
5. Non-smoker (all substances).
6. Specific IgE to HDM (Dermatophagoides farinae) ≥ class 2 in radioallergosorbent test (RAST).
7. BHR (i.e., a decrease in FEV1 of at least 20%) measured by methacholine challenge.
8. FEV1 ≥ 75% of predicted value (according to height, weight and sex).
9. Subject must demonstrate a significant EAR and LAR without rescue medication use within the first 7 hours after BAP.
10. No clinically relevant abnormalities in 12-lead ECG at screening.

Exclusion Criteria:

1. Severe, unstable bronchial asthma.
2. Exacerbation of asthma ≤ 4 weeks prior to screening.
3. Treatment with parenteral and oral corticosteroids 6 weeks prior to screening and during the study.
4. Treatment with inhaled corticosteroids, methylxanthines (e.g., theophyllin), anticholinergics (e.g., ipratropium bromide), leukotriene modifiers (e.g., montelukast), tiotropium bromide, cromolyn or nedocromil within 2 weeks prior to screening and during the study.
5. Current treatment with any immunosuppressants (e.g., monoclonal antibodies, methotrexate, cyclosporin).
6. Specific immunotherapy (SCIT) to mite within 3 years prior to screening.
7. Serious adverse drug reaction to previous biological treatment.
8. Previous therapy with a mAb targeting CD4, including tregalizumab.
9. Known hypersensitivity to any constituents of tregalizumab and/or other mAbs, that, in the opinion of the investigator or Medical Monitor, contraindicates participation.
10. Previous inclusion in this study.
11. Serum transaminases, ALAT and/or ASAT > 2.5-fold ULN at screening.
12. Bilirubin > 34.2 µmol/L at screening.
13. AP > 2-fold ULN at screening.
14. Urea nitrogen > 1.5-fold ULN at screening.
15. Kidney insufficiency as defined by creatinine level > 133 µmol/L at screening.
16. History of severe allergic or anaphylactic reaction to proteins of human origin (e.g. vaccination reaction, biological therapy).
17. Presence or history of malignancy within the previous 5 years (except completely resected squamous or basal cell carcinoma of the skin).
18. Presence or history of clinically significant major disease (e.g., severe heart/lung disease New York Heart Association [NYHA] Class ≥ 3, autoimmune disease [apart from rheumatoid arthritis], acute uncontrolled hyper- or hypo-thyroidism, severe uncontrolled hypo or hypertension).
19. Serious local (e.g., abscess) or systemic (e.g., pneumonia, septicemia) infection or recurrent chronic infections within 6 weeks prior to screening visit or during the screening period.
20. Any infection requiring antibiotic therapy by any route of administration within 4 weeks prior to screening.
21. Vaccination with live, live attenuated, and/or killed vaccines in the 12 weeks prior to the first administration of the study drug and during the study.
22. Positive diagnosis for acute or chronic infections (e.g. HCV, HBV, HIV) at screening or history of previous chronic infection.
23. Acute or clinically symptomatic EBV (infectious mononucleosis) or CMV infection.
24. Presence or history of latent or active tuberculosis.
25. Known immune deficiency.
26. Presence or history of lymphoproliferative disease, including lymphoma and lymphadenopathy.
27. Presence or history of clinically significant drug or alcohol abuse.
28. Employee at study site or any institution involved in this study (including the sponsor), or spouse/partner or relative of an investigator.
29. Pregnant or nursing woman or woman considering to become pregnant during the study or in the 3 months after the last administration of study drug.
30. Woman of childbearing potential (unless surgically sterile or post-menopausal > 52 weeks) who is not using two (2) independent effective contraceptive methods (e.g., oral or injectable contraceptives, intra-uterine devices, double barrier method, contraceptive patch or female sterilization) during the study and for at least 3 months after the last administration of study drug OR Non-vasectomized man who, during the study or in the 3 months after the last administration of study drug, is not using two (2) independent effective contraceptive methods (as specified above) or is planning a sperm donation.
31. Donation of blood within 30 days prior to screening until end of study.
32. Participation in another clinical trial within 90 days before screening or during the study.
33. Inability or lacking motivation to adhere to the study requirements and to comply with the study schedule.
34. Imprisonment or placement in an institution (AMG § 40 (1), sentence 4).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Baseline-corrected late asthmatic response measured by the area under the curve for the forced expiratory volume (FEV1) at 4 to 7 hours after bronchial allergen provocation | Day 84

SECONDARY OUTCOMES:
Change in late asthmatic response, as measured from 4 to 7 hours after bronchial allergen provocation by the maximum decrease in the normalized forced expiratory volume (FEV1) values | Baseline and Day 84
Change in early asthmatic response, as measured from 0 to 3 hours after bronchial allergen provocation by the maximum decrease in the normalized forced expiratory volume (FEV1) values | Baseline and Day 84
Change in early asthmatic response, as measured from 0 to 3 hours after bronchial allergen provocation by the area under the curve of the normalized forced expiratory volume (FEV1) values | Baseline and Day 84
Fraction of eNO (FeNO) absolute levels and delta increase after bronchial allergen provocation | Baseline and Day 84
Dose of methacholine causing a decrease in forced expiratory volume (FEV1) of at least 20% (PD20) | Baseline, Day 85, Day 112
Impact of tregalizumab on TH1, TH2 and TH17 cytokines in blood | Baseline, Day 1, Day 85
Impact of tregalizumab on TH1, TH2 and TH17 cytokines and T-cell transcription factors in sputum | Day 1 until Day 85
Number of eosinophils, neutrophils, macrophages and lymphocytes in sputum | Day 1 until Day 85
Eosinophil cationic protein (ECP) concentration in sputum | Day 1 until Day 85
Number of eosinophils in blood | Baseline, at Day 1, Day 84 and Day 85
Change in mite-specific IgE, IgG4, total IgE and IgG levels in blood | Baseline and Day 84
Impact of tregalizumab on the expression of markers of PBMC lineage in blood | Baseline until Day 112
Incidence and severity of adverse events (AEs) in the participants | Approximatively 27 weeks (study duration)
Levels of specific anti-tregalizumab antibodies in blood | Day 1, Day 36, Day 84
Number of rescue ß2-agonist puffs used | Approximatively for 27 weeks
Change of VAS Nasal Symptom Score | Baseline and Day 84
Quality of life assessed with Asthma Control Test (ACT) and Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12) | Baseline and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — Medaimun GmbH
Locations (1):
- Medaimun GmbH, Frankfurt, Germany